CLINICAL TRIAL: NCT06386536
Title: Cycling for Improved Health: Development and Evaluation of TRIVEL's Smart Bike Training Prescription Programs
Brief Title: Development and Evaluation of TRIVEL Smart Bike Training Prescription Programs.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sylvie Nadeau (Other)
Responsible Party: Sponsor-Investigator, Sylvie Nadeau, Professor, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Organization: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-1796
Record Dates: First submitted 2024-02-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Aging; Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: A single-subject reversal study design (A-B) will be used. During the A and B phases, the participants will undergo training with either the VI-TRIVEL or a conventional stationary bike.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental AB group (Experimental): In this arm, 5 participants will train on the intelligent bike for 5 sessions followed by 5 sessions on a conventional bike (5 participants).
  Interventions: Device: Intelligent stationary bike; Device: Conventional stationary bilke
- Active comparator BA group (Active Comparator): The participants in this arm will start training on a conventional bike for 5 sessions followed by 5 sessions on the intelligent bike (5 participants).
  Interventions: Device: Intelligent stationary bike; Device: Conventional stationary bilke

INTERVENTIONS:
Device: Intelligent stationary bike — A stationary motorized bike prototype that can evaluate lower limb functions such as strength, coordination, range of motion, and tonus. Based on the evaluation results, the iBike proposes a training program that is specific to each individual needs. Moreover, the intelligent bike offers diverse pedaling modes such as forward and backward pedaling, assisted pedaling, isotonic pedaling and pedaling with sensory stimulations.
Device: Conventional stationary bilke — A conventional stationary bike that can be found in gyms or rehab centers.

SUMMARY:
This pilot A-B study aims to develop and validate personalized training programs for older adults with decreased mobility on a Semi-Reclining Intelligent Stationary Bike prototype.

The study also aims to assess the feasibility and acceptability of the training programs and to document their preliminary effects on physical health, perceived well-being, and quality of life. Ten participants will take part in five personalized training sessions with the intelligent bike and five standard training sessions with a traditional stationary bike.

DETAILED DESCRIPTION:
An intelligent stationary bike prototype (iBike) is being developed to evaluate the lower limbs' function during pedaling. The iBike uses artificial intelligence to prescribe personalized training programs based on individual pedaling data. This pilot study aims to develop the training programs, validate their prescription by the iBike, and assess their feasibility, acceptability, and preliminary effects on physical health, perceived well-being, and quality of life in older adults with decreased mobility.

First, the iBike training modules will be developed through a thorough literature review, and prescription criteria will be identified based on the users' pedaling and clinical data as well as expert opinion. Second, 10 participants' lower limb function (i.e. strength, range of motion, coordination and endurance) will be evaluated by the iBike during active and passive pedaling. The evaluation results will be used by the iBike to prescribe a personalized training program. Expert clinicians will also be provided with the ibike evaluation data and will be asked to recommend a personalized exercise program for each participant based on their data. The iBike's prescription of training programs will be validated by comparing it with that of expert clinicians. Third, the feasibility, acceptability, and preliminary effects of the iBike training programs on mobility, physical health, perceived well-being, and quality of life will be assessed through ten training sessions (twice weekly for 45 minutes) with ten older adults using an A-B study design. During the A and B phases, participants will undergo training with either the iBike or a conventional stationary bike.

Ultimately, the goal is to deploy and test this technology in various living spaces and rehabilitation environments to demonstrate its benefits on the physical activity level of healthy older adults and those with mobility problems.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 50 and over
* Having impaired standing mobility associated with aging and/or a stable chronic illness (> 6 months; controlled health condition, no change in medication, routine medical follow-up ; no emergency consultation episode).
* Being able to walk without human assistance for short distances
* Being able to tolerate 90 minutes of activities with rest.
* Being able able to come to the research center for 13 visits, twice a week.

Exclusion Criteria:

* Individuals with or at high risk of having a heart or lung condition (thoracic surgery, angina, myocardial infarction, uncontrolled high blood pressure, shortness of breath at rest).
* Being unable to pedal on a seated stationary bike.
* Having active treatments, including physiotherapy and occupational therapy.
* Having moderate and severe cognitive problems (Mini-Mental State Examination (MMSE) score≤ 21/30).

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Walking ability and functional capacity | 8 to 10 weeks
  2min walk test (2MWT): the participants will be asked to walk as fast as they can, safely, without assistance for two minutes. This outcome will be measured 3 times at baseline and once at the end of each phase of the trial.
Leg strength and endurance | 8-9 weeks
  The sit to stand test: evaluated as the number of stands a person can complete in 30 seconds. This outcome will be measured 3 times at baseline and once at the end of each phase of the trial.

SECONDARY OUTCOMES:
Well-being | 8-9 weeks
  Well being will be assessed with the World Health Organization Well being Index (WHO-5). This outcome will be measured at baseline and at the end of each phase of the trial. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible perception of well being.
Quality of life | 8-9 weeks
  Quality of life will be assessed with the EuroQol Group 5-Dimensions Health Status Questionnaire (EQ5D). This outcome will be measured at baseline and at the end of each phase of the trial.The raw score ranges from 1 to 25, 1 representing best possible and 25 representing worst possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Nadeau, PhD, Principal Investigator — Université de Montréal
Locations (1):
- L'Institut de réadaptation Gingras-Lindsay-de-Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No